CLINICAL TRIAL: NCT05656885
Title: Clinical Evaluation of Proclear Monthly and Avaira Vitality
Brief Title: Clinical Evaluation of Two Frequent Replacement Soft Spherical Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-142
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2022-12

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Intervention Model Description: All participants received Lens A and then Lens B in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): All participants wore Lens A for 15 minutes (Period 1)
  Interventions: Device: Lens A
- Lens B (Experimental): All participants wore Lens B for 15 minutes (Period 2)
  Interventions: Device: Lens B

INTERVENTIONS:
Device: Lens A — Soft spherical hydrogel contact lens for 15 minutes
  Arms: Lens A
Device: Lens B — Soft spherical silicone hydrogel contact lens for 15 minutes
  Arms: Lens B

SUMMARY:
This was a single-blind (participant masked), interventional, prospective, direct refit, bilateral wear short-term fitting study.

DETAILED DESCRIPTION:
The aim of this non-dispensing fitting study was to evaluate the short-term clinical performance of two soft spherical contact lenses after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and signed an information consent letter.
* Self-reports having a full eye examination in the previous two years.
* Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Habitual soft contact lens wearers who currently wear sphere contact lenses, or use spectacles for all distances vision correction, for the past 3 months minimum.
* Has refractive astigmatism no higher than -0.75DC.
* Can be fit and achieve binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deem to be 'acceptable', with the available study lens parameters (powers +8.00 to -12.00DS)

Exclusion Criteria:

* Is participating in any concurrent clinical or research study.
* Has any known active ocular disease and/or infection that contraindicates contact lens wear.
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable.
* Has known sensitivity to the diagnostic sodium fluorescein used in the study.
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment.
* Has undergone refractive error surgery or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan G Carracedo Rodríguez, OD,MSc,PhD, Principal Investigator — University Complutense of Madrid
Locations (1):
- University Complutense of Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens A (Hydrogel Contact Lens): All participants wore Lens A for 15 minutes (Period 1)
- Lens B (Silicone Hydrogel Contact Lens): All participants wore Lens B for 15 minutes (Period 2)
Period: Period 1: Lens A, 15 Minutes
Arm/Group | Lens A (Hydrogel Contact Lens) | Lens B (Silicone Hydrogel Contact Lens)
Started | 40 | 0 (All participants wore Lens A in Period 1)
Completed | 40 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B, 15 Minutes
Arm/Group | Lens A (Hydrogel Contact Lens) | Lens B (Silicone Hydrogel Contact Lens)
Started | 0 (All participants wore Lens B in Period 2) | 40
Completed | 0 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who enrolled and completed all study visits.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.68 (4.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit Acceptance Rating
Description: Measured on lens fit alone on a scale of 0-4 (0=Should not be used; 1=Limit, but unacceptable; 2=Minimum acceptable, early review; 3=Not perfect, but OK to dispense; 4=Perfect) as assessed by an investigator.
Time Frame: 15 minutes
Population: All participants received Lens A and Lens B in sequential order.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens A: All participants that wore Lens A
- Lens B: All participants that wore Lens B
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 40 | 40
score on a scale | 3.28 (0.60) | 3.48 (0.60)

ADVERSE EVENTS:
Time Frame: From dispense up to 15 minutes on each lens type, approximately 1.5 hours.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT05656885/Prot_SAP_000.pdf